CLINICAL TRIAL: NCT05178225
Title: Spa Rehabilitation, Antioxidant and Bioenergetic Supportive Treatment of Patients With Post-Covid-19 Syndrome
Acronym: SpaCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Comenius University (Other)
Collaborators: Sanatórium of Dr. Guhr, n.o. (Unknown); Kaneka Pharma Europe N.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: COVID-19-SK001/2021
Record Dates: First submitted 2022-01-03; First posted 2022-01-05 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: COVID-19 Respiratory Infection
Keywords: Mountain spa rehabilitation; post-COVID-19 syndrome; SARS-CoV-2; pulmonary function; clinical symptoms; platelet mitochondrial metabolism; coenzyme Q10; oxidative stress
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — ubiquinol; ubiquinol-10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patients with post-COVID-19 syndrome with Mountain spa rehabilitation (Active Comparator): patients with post-COVID-19 syndrome with Mountain spa rehabilitation: 15 patients with post-COVID-19 syndrome, 3-6 months after hospitalization were on Mountain spa rehabilitation (MR) in High Tatras, Tatranská Polianka, Slovakia, for 16 to 18 days
  Interventions: Other: mountain spa rehabilitation; Diagnostic Test: 2x14 ml of peripheral blood collected in a tube with anticoagulant
- patients with post-COVID-19 syndrome with Mountain spa rehabilitation + supplementation coenzyme Q10 (Active Comparator): patients with post-COVID-19 syndrome with Mountain spa rehabilitation: 22 patients with post-COVID-19 syndrome, 3-6 months after hospitalization were on Mountain spa rehabilitation (MR) in High Tatras, Tatranská Polianka, Slovakia, 22 patients who will be on spa rehabilitation and at the same time on supplementation with ubiquinol (reduced coenzyme Q10), in a daily dose of 2x100 mg, for 16 to 18 days
  Interventions: Dietary Supplement: ubiquinol (reduced coenzyme Q10); Other: mountain spa rehabilitation; Diagnostic Test: 2x14 ml of peripheral blood collected in a tube with anticoagulant
- healthy control (Placebo Comparator): 15 healthy control volunteers (no Covid-19 or other pathologies)
  Interventions: Diagnostic Test: 2x14 ml of peripheral blood collected in a tube with anticoagulant

INTERVENTIONS:
Dietary Supplement: ubiquinol (reduced coenzyme Q10) — supplementation with ubiquinol (reduced coenzyme Q10), in a daily dose of 2x100 mg. one morning after breakfast, and second dose after dinner.
  Arms: patients with post-COVID-19 syndrome with Mountain spa rehabilitation + supplementation coenzyme Q10
Other: mountain spa rehabilitation — special spa rehabilitation in the mountain High Tatras; Functional capacity of the lungs (6MWT) at before and after 16-18 days of rehabilitation, Borg scale for dyspnea and oxygen saturation SpO2 (%) were monitored.
  Arms: patients with post-COVID-19 syndrome with Mountain spa rehabilitation; patients with post-COVID-19 syndrome with Mountain spa rehabilitation + supplementation coenzyme Q10
Diagnostic Test: 2x14 ml of peripheral blood collected in a tube with anticoagulant — 2x14 ml of peripheral blood collected in a tube with anticoagulant

SUMMARY:
Our hypothesis - that 21 days of mountain spa rehabilitation with ubiquinol supplementation could to accelerate regeneration of patients with post-COVID-19 syndrome, based on the improving platelet mitochondrial bioenergetic, decreasing of oxidative stress and improving of antioxidants protections of patients with post-COVID-19 syndrome.

DETAILED DESCRIPTION:
The first new coronavirus originated from southeast China in 2003 (SARS - Severe Acute Respiratory Syndrome), and the second was originated from Middle East in 2012 (MERS - Middle East Respiratory Syndrome). In March 2020, the World Health Organization declared a global pandemic caused by the SARS-CoV-2 beta-coronavirus responsible for a new type of acute respiratory infection and atypical pneumonia. Persisting signs or symptoms over 12 weeks after the SARS-CoV-2 infection, are defined as post-COVID-19 syndrome. The main symptoms include shortness of breath, general fatigue, exhaustion, headaches, muscle and joint pain, cough, hair, taste and smell loss, sleep and memory disturbances, depression, sensitivity to sound and light.

SARS-CoV-2 viral infection occurs with higher incidence in patients with comorbidities such as diabetes mellitus Type 2, obesity, cardiovascular disease, chronic lung disease and cancer. In aged individuals immune system and mitochondrial dysfunction are a key factors in COVID-19 disease. Mechanical oxygen saturation is required primarily in patients with comorbidities and post-hospitalization pulmonary rehabilitation may be considered in all patients with COVID-19.

Many viruses modulate mitochondrial function, producing more reactive oxygen species, (ROS), cytokine storm, and stimulate inflammation. The investigators published the hypothesis that a target of the new SARS-CoV-2 virus could be mitochondrial bioenergetics and endogenous coenzyme Q10 level. Currently our question was partially answered by authors, who showed reduced mitochondrial bioenergetics in monocytes and peripheral blood mononuclear cells of patients with COVID-19, and the investigators found reduced platelet mitochondrial function in non-hospitalized patients after acute COVID-19 . In the last years isolated platelets from circulating blood are used for estimation of mitochondrial bioenergetics in various diseases, as in patients with chronic kidney diseases, in patients after kidney transplantation, in patients with rheumatoid arthritis. However, the effect of SARS-CoV-2 on platelet mitochondrial function in patients non-vaccinated, hospitalized after infection of SARS-CoV-2 (with post-COVID-19 syndrome), as well as effect of mountain spa rehabilitation on platelet mitochondrial function of patients with post-COVID-19 syndrome has not been published.

Mountain spa rehabilitation (MR) is beneficial for chronic pulmonary diseases, improving fatique, joint pain, psychological stress, sleep disorders and quality of life in patients with various diseases. The investigators assume that special spa rehabilitation in the mountain High Tatras may regenerate impaired mitochondrial metabolism of patients with post-COVID-19 syndrome, can improve physical and mental activity, immunity, reduce oxidative stress and contribute to the acceleration of recovery of patients with post-COVID-19 syndrome.

ELIGIBILITY:
Inclusion Criteria:

* patients with post-COVID-19 syndrome, 3-6 months after hospitalization

Exclusion Criteria:

* no COVID-19 patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
blood count and metabolites | 3 weeks
  2x14 ml of peripheral blood collected in a tube with anticoagulant- two collections before and after Mountain spa rehabilitation Blood count WBC (10to9/L) RBC (10to9/L) HCT (ratio) PLT (10to9/L) MCV (fL) MCH (pg) MCHC (g/L) HgB (g/L)
  Lipids parameters CHOL (mmol/L) HDL-CH (mmol/L) LDL-CH (mmol/L) TAG (mmol/L)
  CRP (mg/L)
lungs function | 3 weeks
  Effect of MR on lungs function Functional capacity of the lungs- walking distance during the 6MWT (m) Exercise dyspnea measured by Borg scale BS (number) Oxygen saturation SpO2 (%)
clinical symptoms (before and after MR) | 3 weeks
  Dry cough Breathing Breathing difficulty Shortness of breath in rest Elevated temperature Chills Heart palpitations Respiratory support with Q2 Weakness Overall fatigue Malaise GIT problems Diarrhea Chest pain Muscle and joint pain Back pain Headache Loss of taste and smell Weight loss Hearing impairment Visual disturbance
damaged platelet mitochondrial bioenergetics | 3 weeks
  Basal oxygen consumption rate in intact platelets (ce) rate of mitochondrial LEAK respiration with CI-linked substrates (1PM - state 4) CI-linked respiration coupled with ATP production (2D- CI-linked oxidative phosphorylation capacity) respiration after addition of cytochrome c (2c) Maximal mitochondrial oxidative capacity (the electron transfer capacity, ET) after uncoupler titration (3U) After addition of exogenous substrate glutamate (4G) non-coupled mitochondrial oxygen consumption Non-coupled oxygen consumption with CI&II-linked substrates (5S) mean of improvement of mitochondrial parameters representing OXPHOS- and electron transport capacity (ET-capacity)
Endogenous coenzyme Q10 and TBARS | 3 weeks
  Endogenous concentration of CoQ10-TOTAL (ubiquinone + ubiquinol) in platelets
  CoQ10-TOTAL in:
  Platelets (pmol.10-9 cells) Blood (µmol.L-1) Plasma (µmol.L-1) TBARS in plasma (µmol.L-1)

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmacobiochemical Laboratory of Third Department of Internal Medicine, Faculty of Medicine Comenius University in Bratislava, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kucharska J, Gvozdjakova A, Mizera S, Braunova Z, Schreinerova Z, Schramekova E, Pechan I, Fabian J. Participation of coenzyme Q10 in the rejection development of the transplanted heart: a clinical study. Physiol Res. 1998;47(6):399-404. PMID 10453746
- [Result] Hilgenfeld R, Peiris M. From SARS to MERS: 10 years of research on highly pathogenic human coronaviruses. Antiviral Res. 2013 Oct;100(1):286-95. doi: 10.1016/j.antiviral.2013.08.015. Epub 2013 Sep 6. PMID 24012996
- [Result] Zhang L, Liu Y. Potential interventions for novel coronavirus in China: A systematic review. J Med Virol. 2020 May;92(5):479-490. doi: 10.1002/jmv.25707. Epub 2020 Mar 3. PMID 32052466
- [Result] Shi TT, Yang FY, Liu C, Cao X, Lu J, Zhang XL, Yuan MX, Chen C, Yang JK. Angiotensin-converting enzyme 2 regulates mitochondrial function in pancreatic beta-cells. Biochem Biophys Res Commun. 2018 Jan 1;495(1):860-866. doi: 10.1016/j.bbrc.2017.11.055. Epub 2017 Nov 9. PMID 29128354
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Li JY, You Z, Wang Q, Zhou ZJ, Qiu Y, Luo R, Ge XY. The epidemic of 2019-novel-coronavirus (2019-nCoV) pneumonia and insights for emerging infectious diseases in the future. Microbes Infect. 2020 Mar;22(2):80-85. doi: 10.1016/j.micinf.2020.02.002. Epub 2020 Feb 20. PMID 32087334
- [Result] Lopez-Lluch G. Mitochondrial activity and dynamics changes regarding metabolism in ageing and obesity. Mech Ageing Dev. 2017 Mar;162:108-121. doi: 10.1016/j.mad.2016.12.005. Epub 2016 Dec 16. PMID 27993601
- [Result] Moreno Fernandez-Ayala DJ, Navas P, Lopez-Lluch G. Age-related mitochondrial dysfunction as a key factor in COVID-19 disease. Exp Gerontol. 2020 Dec;142:111147. doi: 10.1016/j.exger.2020.111147. Epub 2020 Nov 7. PMID 33171276
- [Result] Ganji R, Reddy PH. Impact of COVID-19 on Mitochondrial-Based Immunity in Aging and Age-Related Diseases. Front Aging Neurosci. 2021 Jan 12;12:614650. doi: 10.3389/fnagi.2020.614650. eCollection 2020. PMID 33510633
- [Result] Siddiq MAB, Rathore FA, Clegg D, Rasker JJ. Pulmonary Rehabilitation in COVID-19 patients: A scoping review of current practice and its application during the pandemic. Turk J Phys Med Rehabil. 2020 Nov 9;66(4):480-494. doi: 10.5606/tftrd.2020.6889. eCollection 2020 Dec. PMID 33364571
- [Result] Wang TJ, Chau B, Lui M, Lam GT, Lin N, Humbert S. Physical Medicine and Rehabilitation and Pulmonary Rehabilitation for COVID-19. Am J Phys Med Rehabil. 2020 Sep;99(9):769-774. doi: 10.1097/PHM.0000000000001505. PMID 32541352
- [Result] Maccarone MC, Masiero S. Spa therapy interventions for post respiratory rehabilitation in COVID-19 subjects: does the review of recent evidence suggest a role? Environ Sci Pollut Res Int. 2021 Sep;28(33):46063-46066. doi: 10.1007/s11356-021-15443-8. Epub 2021 Jul 17. PMID 34273080
- [Result] Gvozdjakova A, Klauco F, Kucharska J, Sumbalova Z. Is mitochondrial bioenergetics and coenzyme Q10 the target of a virus causing COVID-19? Bratisl Lek Listy. 2020;121(11):775-778. doi: 10.4149/BLL_2020_126. PMID 33164536
- [Result] Gvozdjakova A, Sumbalova Z, Kucharska J, Chladekova A, Rausova Z, Vancova O, Komlosi M, Ulicna O, Mojto V. Platelet mitochondrial bioenergetic analysis in patients with nephropathies and non-communicable diseases: a new method. Bratisl Lek Listy. 2019;120(9):630-635. doi: 10.4149/BLL_2019_104. PMID 31475544
- [Result] Gvozdjakova A, Sumbalova Z, Kucharska J, Szamosova M, Capova L, Rausova Z, Vancova O, Mojto V, Langsjoen P, Palacka P. Platelet mitochondrial respiration and coenzyme Q10 could be used as new diagnostic strategy for mitochondrial dysfunction in rheumatoid diseases. PLoS One. 2021 Sep 28;16(9):e0256135. doi: 10.1371/journal.pone.0256135. eCollection 2021. PMID 34582480
- [Derived] Gvozdjakova A, Kucharska J, Rausova Z, Lopez-Lluch G, Navas P, Palacka P, Bartolcicova B, Sumbalova Z. Effect of Vaccination on Platelet Mitochondrial Bioenergy Function of Patients with Post-Acute COVID-19. Viruses. 2023 Apr 28;15(5):1085. doi: 10.3390/v15051085. PMID 37243171
- [Derived] Sumbalova Z, Kucharska J, Rausova Z, Palacka P, Kovalcikova E, Takacsova T, Mojto V, Navas P, Lopez-Lluch G, Gvozdjakova A. Reduced platelet mitochondrial respiration and oxidative phosphorylation in patients with post COVID-19 syndrome are regenerated after spa rehabilitation and targeted ubiquinol therapy. Front Mol Biosci. 2022 Oct 21;9:1016352. doi: 10.3389/fmolb.2022.1016352. eCollection 2022. PMID 36339707